CLINICAL TRIAL: NCT02752919
Title: A Single Dose Study to Evaluate the Exposure-Response Relationship Between Galunisertib (LY2157299) and QT Interval in Healthy Japanese and Non-Japanese Subjects
Brief Title: Study of Galunisertib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16214; H9H-MC-JBEI (Other: Eli Lilly and Company.); 2015-005261-23 (EudraCT Number)
Record Dates: First submitted 2016-04-26; First posted 2016-04-27 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
MeSH Terms: interventions — LY-2157299

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A Galunisertib - 1 tablet (Experimental): Single oral dose of galunisertib in Japanese participants
  Interventions: Drug: Galunisertib
- Part A Galunisertib - 2 tablets (Experimental): Single oral dose of galunisertib in Japanese participants
  Interventions: Drug: Galunisertib
- Part B Galunisertib - 1 tablet (Experimental): Single oral dose of galunisertib in non-Japanese participants
  Interventions: Drug: Galunisertib
- Part B Galunisertib - 2 tablets (Experimental): Single oral dose of galunisertib in non-Japanese participants
  Interventions: Drug: Galunisertib

INTERVENTIONS:
Drug: Galunisertib — Administered orally
  Other Names: LY2157299

SUMMARY:
The study involves a single dose of galunisertib taken by mouth by Japanese participants and non-Japanese participants. The study will evaluate the relationship between the effect of the study drug on the electrical activity of the heart, as measured by electrocardiogram (ECG) and how much of the study drug gets into the blood stream and how long it takes the body to remove it. Ths study will last about 42 days for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy male or female Japanese or non-Japanese participants, as determined by medical history and physical examination.
* Male participants: Must agree to use a reliable method of birth control for 12 weeks after receiving the dose of study drug, OR be at least 6 weeks post-vasectomy with documentation of sperm-free ejaculate.
* Female participants: Women not of child-bearing potential may participate, and include those who are:

  * Infertile due to surgical sterilization; or
  * Postmenopausal.
* All female participants must test negative for pregnancy at screening.
* Have a body mass index (BMI) of 18.5 to 32.0 kilogram per meter square (kg/m²), inclusive at screening.
* Have clinical laboratory test results within normal reference range.
* Are able and willing to give signed informed consent.

Exclusion Criteria:

* Have participated, within the last 3 months, in a clinical trial involving an Investigational Product (IP). If the previous IP has a long half-life, 3 months should have passed.
* Have known allergies to galunisertib-related compounds or any components of the formulation, or history of significant atopy.
* Have a personal or family history of long QT syndrome, heart failure, hypokalemia, or sudden death.
* Have a personal history of unexplained syncope within the last year.
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study or affects or confounds the corrected QT (QTc) analysis (the ECG waveform morphology or rhythm are incompatible with reliable measurement of ECG intervals), or have QTcF greater than (>) 450 milliseconds (msec).
* Have an abnormal blood pressure as determined by the investigator.
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the IP; or of interfering with the interpretation of data.
* Have serum magnesium and potassium values outside of the normal reference range.
* Show evidence of human immunodeficiency virus (HIV) infection, hepatitis C or hepatitis B.
* Intend to use over-the-counter or prescription medication (including herbal medications) within 14 days prior to dosing.
* Have donated blood of more than 500 milliliter (mL) within the last month
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Estimated Change from Baseline in Fridericia-corrected QT Interval (QTcF) by Specific Galunisertib Concentrations | Baseline through 72 hours after administration of study drug

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum Drug Concentration (Cmax) of Galunisertib | Predose through 72 hours after administration of study drug
Pharmacokinetics: Time of Cmax (tmax) of Galunisertib | Predose through 72 hours after administration of study drug
Pharmacokinetics: Area Under the Concentration Versus Time Curve (AUC) of Galunisertib | Predose through 72 hours after administration of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Leeds, West Yorkshire, United Kingdom